CLINICAL TRIAL: NCT04261205
Title: Evaluation of the Efficacy and Tolerance of Plasmapheresis by Double Cascade Filtration in a University Centre
Acronym: DFPPSURV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2017/0M-01
Record Dates: First submitted 2019-11-27; First posted 2020-02-07 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Kidney Failure
Keywords: Chronic hemodialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study is being carried out to evaluate the biological, technical and clinical/biological efficacy of this technique, the practice of which is standardized in the department, in order to evaluate our practices and to improve them if necessary. As part of this study, the investigators will ask all patients scheduled for this procedure to participate in this observational prospective study without changing usual practices.

DETAILED DESCRIPTION:
The objective of the study is to conduct a prospective evaluation of the practice of apheresis by Double Filtration System Cascade system in a university centre in current practice with evaluation of the technical and biological effectiveness as the main objective and clinical and biological tolerance as the secondary objective for all consecutive sessions performed in a university centre over a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years of age I indication for plasmapheresis and hospitalized at Chu de Nimes.

Exclusion Criteria:

Under guardianship or curatorship Refusal to participate

Ages: 19 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years of age who consecutively benefit from plasmapheresis sessions by double cascade filtration system during hospitalization at the University Hospital of Nîmes, within the framework of the usual indications retained in the department for a period of 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Apheresis by DFPP and biological efficiency | over a period of one year
  quantification of the purification carried out (volume)

SECONDARY OUTCOMES:
Clinical side effects | within 1 hour of all session
  catheter dysfunction
Biological side effects | within 1 hour of all session
  Bleeding rate
variation of Hb, platelet and albumin before and after session | within 1 hour of all session
  % of Hb, platelet and albumin

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moranne, MD, PhD, Principal Investigator — CHU Nîmes
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Caremeau, Nîmes, France